CLINICAL TRIAL: NCT02179034
Title: Flavors and E-cigarette Effects in Adolescent Smokers- STUDY 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1307012312
Record Dates: First submitted 2014-06-24; First posted 2014-07-01 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Nicotine Dependence, Other Tobacco Product
Keywords: tobacco; electronic cigarettes; menthol; flavors
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Nicotine; Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tobacco Flavor (Placebo Comparator): In this arm, subjects will receive tobacco flavor- without nicotine (placebo). Participants will then be exposed to 3 levels of a menthol additive in random order: no dose, low dose and high dose.
  Interventions: Other: Low Dose Menthol; Other: High Dose Menthol
- Low Dose Nicotine (Active Comparator): In this arm, subjects will receive a low dose of nicotine (6 mg/ml) added to the tobacco flavor. Participants will then be exposed to 3 levels of a menthol additive in random order: no dose, low dose and high dose.
  Interventions: Drug: Nicotine; Other: Low Dose Menthol; Other: High Dose Menthol
- High Dose Nicotine (Active Comparator): In this arm, subjects will receive a high dose of nicotine (12 mg/ml) added to the tobacco flavor. Participants will then be exposed to 3 levels of a menthol additive in random order: no dose, low dose and high dose.
  Interventions: Drug: Nicotine; Other: Low Dose Menthol; Other: High Dose Menthol

INTERVENTIONS:
Drug: Nicotine — Participants will receive no nicotine, low dose nicotine (6 mg/ml) or high dose nicotine (12 mg/ml)
  Arms: High Dose Nicotine; Low Dose Nicotine
Other: Low Dose Menthol — A low dose of menthol will be added to the tobacco flavor.
Other: High Dose Menthol — A high dose of menthol will be added to the tobacco flavor.

SUMMARY:
This study is to examine if inhaled doses of menthol that produce low and high cooling effects change the appeal of e-cigarettes containing low and high doses of nicotine in adolescent smokers. The hypothesis is that the combination of nicotine and menthol, when compared with menthol or nicotine alone, will result in greater increase in liking of an e-cigarette and greater reduction in nicotine withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-20 years
* Able to read and write
* Cigarette smoker
* Use of e-cigarettes in the past 30 days

Exclusion Criteria:

* Seeking smoking cessation treatment
* Current/lifetime criteria for dependence on another psychoactive substance -Daily use of alcohol or marijuana or use of any other drugs including cocaine, opiates, stimulants
* Regular use of psychoactive drugs including anxiolytics, antidepressants and other psychostimulants
* Current or past history of psychosis or other psychiatric diagnosis such as major depression
* Any significant current medical condition

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2016-07-18 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Liking/effect score of the e-cigarette | Every 30 min for 120 min during lab session
  The Drug Effects Questionnaire (Soria et al) will be used to ask about participants' liking/effect of the e-cigarettes smoked during the 4 bouts of e-cigarette puffing during the lab session to determine which menthol dose is most preferred. A linear mixed-effects regression model wil be used with nicotine group (none, low, high) as between-subject factor, and menthol dose (none, low dose, high dose) as within-subject factor.

SECONDARY OUTCOMES:
Maximum value of money at which the e-cigarette is chosen over money | Every 30 min for 120 min during lab session
  E-cigarette value will be determined using the Multiple Choice Procedure (Griffiths et al, 1993) to determine the reinforcing value of the e-cigarette. The MCP involves sampling the e-cigarette and then making a discrete choice between the e-cigarette or a series of monetary values.
Change scores from baseline in Nicotine Withdrawal | Every 30 min for 120 min during lab session
  The Minnesota Nicotine Withdrawal Scale (Hughes et al,1986) will be used to assess the magnitude of change in nicotine withdrawal symptoms during the lab session
Change scores from baseline in Tobacco Craving | Every 30 min for 120 min during lab session
  The Brief Questionnaire on Smoking Urges (Tiffany & Drobes,1991) will be used to assess the magnitude of change in tobacco craving during the lab session

CONTACTS AND LOCATIONS:
Overall Officials: Dana Cavallo, PhD, Study Director — Yale University
Locations (1):
- CMHC, New Haven, Connecticut, United States